CLINICAL TRIAL: NCT04811560
Title: A Phase 1/2, First-in-Human Study of the Menin-KMT2A (MLL1) Inhibitor Bleximenib in Participants With Acute Leukemia (cAMeLot-1)
Brief Title: A Phase 1/2 Study of Bleximenib in Participants With Acute Leukemia (cAMeLot-1)
Acronym: cAMeLot-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108998; 75276617ALE1001 (Other: Janssen Research & Development, LLC); 2023-506581-31-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2021-03-22; First posted 2021-03-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Acute Leukemias; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bleximenib (Experimental): Participants in Phase 1 Part 1 (dose escalation) will receive bleximenib orally. The dose levels will be escalated based on the dose limiting toxicities (DLT) evaluation by Study Evaluation Team (SET) until the recommended Phase 2 Doses (RP2Ds) have been identified. Participants in Phase 1 Part 2 (dose expansion) will receive bleximenib orally at the RP2D(s) determined in Part 1. In Phase 2 participants will receive bleximenib at the RP2D to evaluate anti-leukemia activity and demonstrate acceptable safety at the RP2D(s).
  Interventions: Drug: Bleximenib

INTERVENTIONS:
Drug: Bleximenib — Bleximenib is administered orally.
  Other Names: JNJ-75276617

SUMMARY:
The purpose of this study is to determine the recommended Phase 2 dose(s) (RP2D[s]) of bleximenib in phase 1 Part 1 (Dose Escalation) and to determine the safety and tolerability at RP2D in Phase 1 Part 2 (Dose expansion). The purpose of the Phase 2 part of the study is to evaluate the efficacy of bleximenib at the RP2D.

ELIGIBILITY:
Inclusion Criteria:

Phase 1:

* Age 2 years and above (pediatric cohort only), all other cohorts 18 years and above
* Relapsed or refractory (R/R) acute leukemia and has exhausted, or is ineligible for, available therapeutic options
* Acute leukemia harboring histone-lysine N-methyltransferase 2A (KMT2A), nucleophosmin 1 gene (NPM1) or nucleoporin 98 gene or nucleoporin 214 gene (NUP98 or NUP214) alterations

Phase: 2

* Participants greater than 18 years are eligible
* Must have had an initial diagnosis of acute myeloid leukemia (AML) per the WHO 2022 classification criteria and have relapsed/refractory disease
* AML harboring KMT2A-r (gene rearrangement/translocation) or NPM1 mutations only

For Both Phase 1 and 2:

* Pretreatment clinical laboratory values meeting the following criteria: (a) Hematology: white blood cell (WBC) count less than or equal to (<=) 20*10^9/liter (L) and (b) renal function; For adult participants, estimated or measured glomerular filtration rate greater than equal (>=) 30 milliliter per minute (mL/min) per four variable MDRD equation. For pediatric participants an estimated or measured glomerular filtration rate >50 mL/min per the CKiD (Chronic Kidney Disease in Children) Schwartz formula
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0, 1 or 2. Pediatric participants only: Performance status >=70 by Lansky scale (for participants less than [<]16 years of age) or >=70 Karnofsky scale (for participants >=16 years of age)
* A female of childbearing potential must have a negative highly sensitive serum beta-human chorionic gonadotropin at screening and within 48 hours prior to the first dose of study treatment
* Participant must agree to all protocol required contraception requirements and avoid sperm or egg donations or freezing for future reproductive use while on study and for 90 days (males) or 6 months (females) after the last dose of study treatment

Exclusion Criteria:

* Acute promyelocytic leukemia, diagnosis of Down syndrome associated leukemia or juvenile myelomonocytic leukemia according to World Health Organization (WHO) 2016 criteria
* Active central nervous system (CNS) disease
* Prior solid organ transplantation
* QTc according to Fridericia's formula (QTcF) for males >= 450 millisecond (msec) or for females >= 470 msec. Participants with a family history of Long QT syndrome are excluded
* Exclusion criteria related to stem cell transplant: a. Received prior treatment with allogenic bone marrow or stem cell transplant <=3 months before the first dose of study treatment; b. Has evidence of graft versus host disease; c. Received donor lymphocyte infusion <=1 month before the first dose of study treatment; d. Requires immunosuppressant therapy (exception: daily doses <=10 milligrams (mg) prednisone or equivalent are allowed for adrenal replacement)
* Prior cancer immunotherapy within 4 weeks prior to enrollment or blinatumomab within 2 weeks prior to enrollment. Additional prior cancer therapies must not be given within 4 weeks prior to enrollment or 5 half-lives of the agent (whichever is shorter)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2026-02-16 (Estimated); Study Completion 2028-05-26 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 4 years and 9 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Phase 1: Number of Participants with AEs by Severity | Up to 4 years and 9 months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Phase 1: Part 1: Percentage of Participants with Dose-Limiting Toxicity (DLT) | Up to 28 days Cycle 1
  Percentage of participants with DLT will be assessed accordingly to national cancer institute common terminology criteria for adverse events (NCI-CTCAE) version 5.
Phase 2: Rate of Complete Remission or Complete Remission with Partial Hematologic Recovery (CR/CRh) | Up to 4 years and 9 months
  Rate of CR/CRh is defined as the percentage of participants achieving a CR or CRh at any time post-treatment.

SECONDARY OUTCOMES:
Phase 1 and 2: Plasma Concentration of Bleximenib | Up to 4 years and 9 months
  Plasma concentration of bleximenib will be reported.
Phase 1 and 2: Overall Response Rate (ORR) | Up to 4 years and 9 months
  ORR is defined as the percentage of participants who achieve any response.
Phase 1: Duration of Response (DOR) | Up to 4 years and 9 months
  DOR will be calculated among responders from the date of initial documentation of a response to the date of first documented evidence of relapse, as defined in the disease-specific response criteria, or death due to any cause, whichever occurs first.
Phase 1 and 2: Time To Response (TTR) | Up to 4 years and 9 months
  TTR is defined for the responders as the time from the date of the first dose of bleximenib to the date of the first documented response.
Phase 2: Duration of Complete Response (CR)/Complete Remission With Partial Hematologic Recovery (CRh) | Up to 4 years and 9 months
  The duration of CR/CRh is defined from the date of first CR or CRh response achieved to the date of first evidence of relapsed disease or death due to any cause, whichever occurs first, for participants who achieve a CR or CRh.
Phase 2: Time To CR/CRh | Up to 4 years and 9 months
  Time to CR/CRh is defined for responders as the time from the date of the first dose of bleximenib to the date of first achieving either CR or CRh, depending on which milestone is reached.
Phase 2: Event-free survival (EFS) | Up to 4 years and 9 months
  EFS is defined as the time from the date of first dose of study treatment to the date of treatment failure, relapse, or death due to any cause, whichever occurs first.
Phase 2: Overall survival (OS) | Up to 4 years and 9 months
  OS is defined from the date of first dose of study treatment to the date of death due to any cause.
Phase 2: Measurable Residual Disease (MRD) Negativity Among Participants Achieving CR/CRh/CRi | Up to 4 years and 9 months
  MRD-negative rate is defined as the percentage of participants who are MRD-negative at any timepoint after the first dose of bleximenib in the responders.
Phase 2: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 4 years and 9 months
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. A Serious AE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Phase 2: Number of Participants Reporting Transfusion Independence | Up to 4 years and 9 months
  Transfusion independence is defined as independence from red blood cells (RBC) and platelet transfusions during any 56-day interval after receiving study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (101):
- United States (27):
  - City of Hope Phoenix, Goodyear, Arizona
  - City of Hope, Duarte, California
  - University of California Irvine Medical Center, Orange, California
  - University of California San Francisco, San Francisco, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - University of Chicago, Chicago, Illinois
  - St Francis Hospital & Health Centers Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Start Midwest, Grand Rapids, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - NYU Langone Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Oregon Health And Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Maine Health, Providence, Rhode Island
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - MD Anderson, Houston, Texas
  - San Antonio Methodist TX Transplant Physicians Group, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Medical College of WI at Froedtert, Milwaukee, Wisconsin
- Australia (3):
  - Monash Medical Centre, Clayton
  - Royal Perth Hospital, Perth
  - Gold Coast University Hospital, Southport
- Brazil (6):
  - Instituto D Or de Pesquisa e Ensino, Brasília
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Ministerio da Saude Instituto Nacional do Cancer, Rio de Janeiro
  - Fundacao Faculdade de Medicina Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Instituto D Or de Pesquisa e Ensino IDOR, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
- Canada (3):
  - Vancouver Coastal Health, Vancouver, British Columbia
  - Princess Margaret Cancer Centre University Health Network, Toronto, Ontario
  - Hopital Maisonneuve Rosemont, Montreal, Quebec
- China (12):
  - Peking University First Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - West China Hospital Si Chuan University, Chengdu
  - Nanfang Hospital of Southern Medical Hospital, Guangzhou
  - First Affiliated Hospital Medical School of Zhejiang University, Hangzhou
  - Qilu Hospital of Shandong University, Jinan
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Zhongda Hospital Southeast University, Nanjing
  - Institute of Hematology and Blood Diseases Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - Henan Cancer Hospital, Zhengzhou
- France (13):
  - Hopital Jean Minjoz, Besançon
  - Institut Paoli Calmettes, Marseille
  - CHU de Nantes hotel Dieu, Nantes
  - Hopital Saint Louis, Paris
  - Hopital trousseau- APHP, Paris
  - Centre Hospitalier Universitaire (CHU) de Bordeaux Hopital HautLeveque Centre Francois Magendie, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - Institut de Cancerologie Strasbourg Europe ICANS, Strasbourg
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - CHU Bretonneau, Tours
  - CHRU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy
  - CHRU Nancy Brabois, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Israel (4):
  - Carmel Medical Center, Haifa
  - Hadassah University Hospita Ein Kerem, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Japan (11):
  - Kyushu University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Kanazawa University Hospital, Kanazawa
  - National Cancer Center Hospital East, Kashiwa
  - Kobe City Medical Center General Hospital, Kobe
  - Gunmaken Saiseikai Maebashi Hospital, Maebashi
  - Nagoya University Hospital, Nagoya
  - Hokkaido University Hospital, Sapporo
  - NTT Medical Center Tokyo, Tokyo
  - Yamagata University Hospital, Yamagata
  - University of Fukui Hospital, Yoshida
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Clinico Univ. de Valencia, Valencia
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (8):
  - University Hospital of Wales, Cardiff
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - The Clatterbridge Cancer Centre, Liverpool
  - Guys and St Thomas NHS Foundation Trust, London
  - University College London Hospitals, London
  - The Christie Nhs Foundation Trust, Manchester
  - Oxford University Hospitals NHS Trust, Oxfordshire
  - University Hospitals Plymouth NHS Trust, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Kwon MC, Thuring JW, Querolle O, Dai X, Verhulst T, Pande V, Marien A, Goffin D, Wenge DV, Yue H, Cutler JA, Jin C, Perner F, Hogeling SM, Shaffer PL, Jacobs F, Vinken P, Cai W, Keersmaekers V, Eyassu F, Bhogal B, Verstraeten K, El Ashkar S, Perry JA, Jayaguru P, Barreyro L, Kuchnio A, Darville N, Krosky D, Urbanietz G, Verbist B, Edwards JP, Cowley GS, Kirkpatrick R, Steele R, Ferrante L, Guttke C, Daskalakis N, Pietsch EC, Wilson DM, Attar R, Elsayed Y, Fischer ES, Schuringa JJ, Armstrong SA, Packman K, Philippar U. Preclinical efficacy of the potent, selective menin-KMT2A inhibitor JNJ-75276617 (bleximenib) in KMT2A- and NPM1-altered leukemias. Blood. 2024 Sep 12;144(11):1206-1220. doi: 10.1182/blood.2023022480. PMID 38905635